CLINICAL TRIAL: NCT05388890
Title: Clinical Study on the Efficacy of Modified Liujunzi Prescription on the Treatment of Atrophic Gastritis After HP Eradication
Brief Title: Treatment of Atrophic Gastritis After HP Eradication With Modified Liujunzi Decoction Based on Syndrome Differentiation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShouFa-2022-2-4077
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Chronic Atrophic Gastritis
Keywords: Chronic Atrophic Gastritis; Modified Liujunzi Decoction; Treatment Based on Syndrome Differentiation; Clinical Study; Efficacy; Cohort Study
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood;Biopsy specimen of gastric mucosa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MLD: Modified Liujunzi Decoction,1 package twice daily,6 months
  Interventions: Drug: MLD
- WFC: Weifuchun,three times a day, four at a time,6months
  Interventions: Drug: WFC

INTERVENTIONS:
Drug: MLD — Modified Liujunzi Decoction is provided by the chinese pharmacy of Peking University First Hospital , one dose per day, taken in twice, and the course of treatment is 6 months.
  Groups: MLD
Drug: WFC — Chinese patent medicine, take according to the instructions, the course of treatment is 6 months.
  Groups: WFC

SUMMARY:
This is an observational cohort study of clinical efficacy study.The purpose of this topic is to evaluate the efficacy and safety of Modified Liujunzi Decoction based on syndrome differentiation in patients with chronic atrophic gastritis(CAG) after HP eradication.Taking Modified Liujunzi Decoction as the observation group and Weifuchun routine treatment as the control group, so as to provide evidence for the treatment of CAG and reduce the risk of gastric cancer. A total of 284 patients were included. The curative efficacy, symptom score and adverse events will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CAG diagnosed by endoscopy and pathological examination, the pathological diagnosis criteria refer to the China consensus of chronic gastritis (2017) ;
* Previous HP infection, HP negative after standardized treatment;
* TCM syndrome differentiation mainly focuses on the weakness of the spleen and stomach,referring to the consensus on the diagnosis and treatment of chronic atrophic gastritis with integrated traditional Chinese and Western Medicine (2017), there is no restriction on concurrent syndrome;
* Age 18-70 years old, regardless of gender;
* The subject (or legal representative) voluntarily agreed and signed the informed consent form, and was able to abide by the study protocol during the study.

Exclusion Criteria:

* History of gastric surgery;
* Combined with serious diseases affecting the study evaluation, such as serious liver disease, heart disease, kidney disease, malignant tumor and alcoholism;
* Allergic to the drugs used in this study;
* Participated in clinical research of other drugs in the first 3 months of the study;
* Patients can't express correctly their subjective feelings and can't cooperate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the willingness of the patients, the CAG patients after HP eradication in the routine diagnosis and treatment of the Department of integrated traditional Chinese and Western medicine and the Department of Gastroenterology of the Peking University First Hospital were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapeutic effectiveness of gastric mucosal lesions | Half a year,a year
  Referring to the CAG of the "Guidelines for Clinical Research on New Chinese Medicines (2002)", the effective treatment of gastric mucosal lesions is defined as "the pathological score decreased by 1 point compared with the previous point". The effective rate of gastric mucosal lesions treatment = the number of cases with a decrease of ≥ 1 point by the previous score / the total number of cases × 100%. The effective rate of gastric mucosal lesions from different category will be calculated: respectively for atrophy, chronic inflammation, activity, intestinal metaplasia, and intraepithelial neoplasia .

SECONDARY OUTCOMES:
The efficacy of OLGA,OLGIM | Half a year,a year
  The efficacy of OLGA staging: OLGA staging decreased by ≥1 stage compared with the baseline is considered as effecacy.The effective rate = the number of cases with ≥1 stage decreased compared with the previous stage/the total number of cases × 100%.
  The efficacy of OLGIM staging:The OLGIM staging decreased by ≥1 stage from the baseline is considered effective for patients with intestinal metaplasia. The effective rate = the number of cases staging decreased by ≥ 1 stage compared with the previous stage /the total number of cases × 100%
Changes in clinical symptom scores | The third month,half a year ,the ninth month,a year.
  Evaluate referring to the symptom grading and quantification standard of "Guidelines for Clinical Research on Chronic Atrophic Gastritis" from "Guidelines for Clinical Research on New Chinese Medicines (2002)".According to the clinical symptom severity assign different points. No, mild, moderate and severe symptoms are recorded as 0, 1, 2, and 3 point respectively. Record the changes of the symptom score at 6 months and 12 months compared with the baseline and evaluate . The calculation formula is " the total score after treatment-the score in baseline ".
The recurrence of HP | Half a year,a year
  13C-UBT was performed to determine HP, and the DOB value more than 4 is defined as the recurrence of HP.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided